CLINICAL TRIAL: NCT07183826
Title: Internet-Based Mindfulness-Based Cognitive Therapy (iMBCT) for Chronic Tinnitus Patients: a Randomized Controlled Trial Protocol
Brief Title: Internet-Based Mindfulness-Based Cognitive Therapy (iMBCT) for Chronic Tinnitus Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warsaw (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Paweł Holas, MD, PhD, associate professor, University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8/04/2023
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Tinnitus; Anxiety; Depressive
Keywords: chronic tinnitus; tinnitus; Mindfulness-Based Cognitive Therapy; MBCT; Internet-delivered intervention; Online mental health; Depression; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Tinnitus; Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: This study used a two-arm, parallel-group randomized controlled trial design. Participants meeting inclusion criteria were randomly assigned to one of two conditions: (1) unguided internet-delivered Mindfulness-Based Cognitive Therapy (iMBCT), or (2) a waitlist control (WLC). Randomization was stratified by demographic characteristics and baseline symptom severity to ensure balanced groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Delivered Mindfulness-Based Cognitive Therapy (iMBCT) (Experimental): A 6-week (42 days), unguided online adaptation of the Mindfulness-Based Cognitive Therapy (MBCT) program. The intervention consisted of six sequential modules delivered through a secure web platform, including guided mindfulness meditations, body scan, mindful movement, and cognitive-behavioral exercises. Participants received audio recordings, written materials, and reflective tasks, along with automated reminder emails. No therapist guidance was provided.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (Internet-delivered)
- Waiting List Control (Placebo Comparator): Participants in this arm received no active intervention during the 6-week waitlist period but completed all study assessments on the same schedule as intervention arms. After the waiting period, participants were offered to take part in the online MBCT program.
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (Internet-delivered) — A 6-week (42 days), unguided online adaptation of the Mindfulness-Based Cognitive Therapy (MBCT) program. The intervention consisted of six sequential modules delivered through a secure web platform, including guided mindfulness meditations, body scan, mindful movement, and cognitive-behavioral exercises. Participants received audio recordings, written materials, and reflective tasks, along with automated reminder emails. No therapist guidance was provided.
  Arms: Internet-Delivered Mindfulness-Based Cognitive Therapy (iMBCT)
Behavioral: No intervention — Participants in this arm received no active intervention during the 6-week waitlist period but completed all study assessments on the same schedule as intervention arms. After the waiting period, participants were offered to take part in the online MBCT program.
  Arms: Waiting List Control

SUMMARY:
This study tested a 6-week, internet-based Mindfulness-Based Cognitive Therapy (MBCT) program designed to help people experiencing distress related to chronic tinnitus. Tinnitus is condition that can cause anxiety, depression, and negatively impact the quality of life.

The investigators compare the online MBCT program to a wait-list group. Study aims to measure tinnitus distress, symptoms of anxiety, depression, mindfulness traits, and self-compassion before the program, right after, one month later, and six months later.

DETAILED DESCRIPTION:
Tinnitus, the perception of sound without an external source, affects about 10-15% of people worldwide, with 2-3% experiencing severe distress. Large studies estimate that around 14% of adults report tinnitus, and about 2% suffer from a disabling form. In Europe, roughly one in seven adults is affected. Tinnitus often occurs alongside anxiety, depression, insomnia, and reduced quality of life. Even mild tinnitus has been linked to poorer sleep and higher levels of anxiety and depression.

Despite extensive research, there is no universal medical cure for tinnitus. As a result, treatment increasingly focuses on psychological and behavioral methods that aim to reduce distress and promote habituation. Cognitive Behavioral Therapy (CBT) is the current gold standard, reliably easing distress and improving coping, though it is not effective for everyone and access remains limited. This has led to growing interest in mindfulness-based approaches, such as Mindfulness-Based Cognitive Therapy (MBCT), which combine mindfulness practices with cognitive strategies focused on acceptance rather than control of symptoms.

Mindfulness-based treatments target the negative thoughts, catastrophic interpretations, and avoidance behaviors that sustain tinnitus distress. Acceptance of tinnitus has been shown to improve quality of life and reduce depression and distress. By fostering non-judgmental awareness of the present moment, MBCT helps patients shift from struggling against tinnitus toward acceptance.

Clinical research shows that mindfulness approaches can reduce tinnitus severity, psychological distress, and negative thinking. Trials demonstrate that MBCT and Mindfulness-Based Stress Reduction (MBSR) are effective, with some studies finding MBCT more beneficial than relaxation therapies, and benefits lasting for months. Online versions of mindfulness-based tinnitus programs have also proven feasible and helpful, particularly during the COVID-19 pandemic. Ongoing studies directly comparing MBCT with CBT further highlight the expanding role of mindfulness in tinnitus care.

Mindfulness-Based Cognitive Therapy (MBCT) MBCT is an eight-week, group-based psychological program originally developed to prevent relapse in recurrent depression. It combines mindfulness meditation practices with cognitive-behavioral therapy strategies, fostering non-judgmental awareness of present-moment experience, greater cognitive flexibility, and reduced reactivity to negative thoughts and emotions.

Mechanistic research suggests that MBCT works by:

Increasing cognitive defusion - the ability to step back from and observe thoughts without automatically believing or reacting to them. Reducing experiential avoidance - the tendency to suppress or avoid difficult emotions and sensations. Enhancing self-compassion - a kinder, more understanding stance toward oneself in times of suffering.

Internet-Delivered MBCT (iMBCT) Internet-delivered psychological interventions (IPIs) have the potential to greatly expand access to evidence-based care. Online MBCT (iMBCT) can be delivered synchronously (live sessions with a facilitator) or asynchronously (self-paced, unguided), with evidence supporting effectiveness in reducing distress and improving resilience. Unguided iMBCT programs are especially promising for public health implementation due to their low delivery cost and scalability, but high-quality trials in specific clinical groups remain rare.

Study Objectives The main objective of the planned research is to evaluate the effectiveness of an iMBCT intervention for tinnitus distress, depression, and anxiety symptoms among chronic tinnitus patients.

More specific objectives are as follows: (1) evaluate the effectiveness of the intervention relative to waiting-list according to self-reported measures; (2) conduct an examination of predictors and mediators of treatment response; (3) evaluate the maintenance of tinnitus distress alleviation as well as anxiety and depression symptoms at 1-month and 6-month follow-up.

Study design and setting This study is a two-arm, parallel-group, randomized controlled trial (RCT) comparing iMBCT with a waiting list control. A CONSORT-compliant flowchart (Figure 1) depicts participant progression. The participants will be allocated to either a 6-week iMBCT intervention, or (2) waiting-list control group (WLC).

Participants will be instructed to contact the research team in the event of a crisis, at which point they will be assessed by a study-affiliated psychotherapist or psychiatrist and referred to appropriate clinical services as necessary.

All assessments will be conducted via an online data collection platform provided by the investigators (terapiawszumach.pl) at the following time points: (1) screening, (2) baseline (prior to randomization), (3) upon completion of the 6-week online program or waitlist period, (4) one month post-treatment (for participants in the active intervention groups), and (5) six months post-treatment.

ELIGIBILITY:
Inclusion criteria

1. Willingness and ability to participate in online therapy.
2. Polish language proficiency.
3. 18 years or older.
4. Suffering from chronic tinnitus for at least 3 months.
5. A score of ≥32 on the TFI. Exclusion criteria

1) Mentally incapable patients. 2) Patients who have already completed structured mindfulness training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Change in Tinnitus Distress | Screening, Baseline (Week 0), Post-intervention (Week 6), Follow-ups (Week 10, 32)
  Change in Tinnitus Distress from baseline to post-intervention, and follow-up, measured by TFI is a 25-item instrument designed to assess the impact of tinnitus on various aspects of daily functioning, using 11-point Likert scales. Total scores range from 0 to 100, with a minimum clinically important difference (MCID) of 13 points and higher scores indicating greater distress.
Anxiety and Depression symptoms | Screening, Baseline (Week 0), Post-intervention (Week 6), Follow-ups (Week 10, 32)
  Instrument: Hospital Anxiety and Depression Scale (HADS), a 14-item self-report instrument designed to assess symptoms of anxiety and depression, with each item rated on a four-point scale. It consists of two sub-scales: HADS-anxiety and HADS-depression, 7 items each. The two-factor structure has been verified. Each sub-scale yields a score ranging from 0 to 21, with higher values indicating more symptoms.

SECONDARY OUTCOMES:
Acceptance of Tinnitus | Screening, Baseline (Week 0), Post-intervention (Week 6), Follow-ups (Week 10, 32)
  Instrument: Tinnitus Acceptance Questionnaire (TAQ), a 12-item questionnaire developed specifically for measuring acceptance in patients with CT. Each item is evaluated on a scale from 0 (never true) to 6 (always true), and their scores are combined to determine a total score, with a maximum of 72 points. Higher scores indicate higher levels of acceptance.
Self-compassion | Screening, Baseline (Week 0), Post-intervention (Week 6), Follow-ups (Week 10, 32)
  Instrument: the Self-Compassion Scale-Short Form (SCS-SF), a 12-item questionnaire developed to assess the capacity for self-compassion. It comprises two sub-scales: self-disparagement and self-care, each consisting of six items. Overall score fall in range 1 to 5 and are the mean value of 12 items after reverse scoring negatively worded items. Higher total scores reflect greater self-compassion, characterized by elevated self-care and reduced self-disparagement.
cognitive and affective mindfulness | Screening, Baseline (Week 0), Post-intervention (Week 6), Follow-ups (Week 10, 32)
  Instrument: Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), a 12-item scale that gauges everyday mindfulness by centering on how respondents encounter their thoughts and emotions. Each item is evaluated on a 4-point Likert scale, ranging from 1 (rarely/not at all) to 4 (almost always). Higher scores indicate heightened levels of mindfulness
Emotion Regulation | Screening, Baseline (Week 0), Post-intervention (Week 6), Follow-ups (Week 10, 32)
  Instrument: The Difficulties in Emotion Regulation Scale (DERS-16), a 16-item assessment tool designed to evaluate difficulties in emotion regulation. Respondents rate items using a 5-point Likert scale, where higher scores indicate greater difficulties in emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Holas, MD, PhD, Study Director — University of Warsaw
Locations (1):
- Faculty of Psychology, University of Warsaw, Warsaw, Poland